CLINICAL TRIAL: NCT00515437
Title: A Multi-Center, Randomized, Double-blind, Placebo-Controlled,Sequential Dose Escalation, Safety, Tolerability, and Preliminary Efficacy Study of MYOBLOC for the Treatment of Sialorrhea in Parkinson's Disease Patients
Brief Title: A Multi-Center Study of MYOBLOC for the Treatment of Sialorrhea in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solstice Neurosciences (Industry)
Responsible Party: Sponsor
Organization: USWM, LLC (dba US WorldMeds) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SN-SIAL-201
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Drooling
Keywords: Sialorrhea
MeSH Terms: conditions — Sialorrhea | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 1500U Myobloc
  Interventions: Biological: Botulinum Toxin Type B (Myobloc)
- 2 (Experimental): 2500U Myobloc
  Interventions: Biological: Botulinum Toxin Type B (Myobloc)
- 3 (Experimental): 3500U Myobloc
  Interventions: Biological: Botulinum Toxin Type B (Myobloc)
- 4 (Placebo Comparator): pooled placebo
  Interventions: Biological: Matched placebo to Myobloc

INTERVENTIONS:
Biological: Botulinum Toxin Type B (Myobloc)
  Arms: 1; 2; 3
Biological: Matched placebo to Myobloc
  Arms: 4

SUMMARY:
To determine safety, tolerability and preliminary efficacy of intraglandular injections of MYOBLOC for the treatment of sialorrhea in Parkinsons' Disease patients

DETAILED DESCRIPTION:
This is a multi-center, outpatient, double-blind, placebo-controlled, single treatment, sequential dose escalation study designed to evaluate the safety, tolerability and preliminary efficacy of single doses of MYOBLOC versus placebo for the treatment of sialorrhea in Parkinson's disease patients, lasting approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Parkinsons' Disease patients with Sialorrhea for at least 3 months

Exclusion Criteria:

* Patients with non-idiopathic PD parkinsonism
* Patients previously exposed to botulinum toxins
* Patients with a history of aspiration pneumonia, moderate/severe choking and/or moderate/severe dysphagia
* Patients with prior salivary gland surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pappert, MD, Study Director — Solstice Neurosciences
Locations (18):
- United States (18):
  - Dr Virgilio Evidente, Scottsdale, Arizona
  - Dr. Ronald Ziman, Northridge, California
  - Dr. James Sutton, Oxnard, California
  - Dr. Olga Klepitskaya, Denver, Colorado
  - Dr. Fernando Pagan, Washington D.C., District of Columbia
  - Dr Hubert Fernandez, Gainesville, Florida
  - Dr. Alan Freeman, Atlanta, Georgia
  - Dr. Katie Kompoliti, Chicago, Illinois
  - Dr. Robert Rodnitzky, Iowa City, Iowa
  - Dr. Stephen Reich, Baltimore, Maryland
  - Dr. Brad Racette, St Louis, Missouri
  - Dr. Eric Molho, Albany, New York
  - Dr. Joseph Friedman, Warwick, Rhode Island
  - Dr. Vanessa Hinson, Charleston, South Carolina
  - Dr. Sam Kabbani, Knoxville, Tennessee
  - Dr. Madhavi Thomas, Dallas, Texas
  - Dr. Gordon Smith, Salt Lake City, Utah
  - Dr. Patrick Hogan, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 centers were initiated to screen and enroll subjects. Enrollment began in July 2007 and completed in March 2008. 54 subjects were enrolled at 17 centers
Groups:
- 1500U Myobloc: 1500U Myobloc
- 2500U Myobloc: 2500U Myobloc
- 3500U Myobloc: 3500U Myobloc
- Placebo: Placebo
Period: Overall Study
Arm/Group | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Started | 14 | 12 | 13 | 15
Completed | 14 | 12 | 13 | 14
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo | Total
Number analyzed (Participants) | 14 | 12 | 13 | 15 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 0 | 3 | 10
  >=65 years | 9 | 10 | 13 | 12 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7) | 71 (8) | 74 (5) | 71 (11) | 71 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 2 | 6
  Male | 12 | 12 | 11 | 13 | 48
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 13 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Drooling Frequency & Severity Scale (DFSS)at Wk 4 Post-injection
Description: 9 point scale, 0 = no drooling, 9 = severe drooling
Time Frame: baseline versus 4 weeks post-injection
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 14
points on a scale | -2.1 (1.2) | -3.3 (1.4) | -3.5 (1.0) | -1.3 (1.3)

2. Secondary Outcome: Change in Drooling Frequency and Severity Scale (DFSS) at Wk 12 Post-injection
Description: 9 point scale (0=no drooling, 9=severe drooling)
Time Frame: baseline vs 12 weeks post injection
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 14
points on a scale | -1.9 (1.5) | -2.2 (1.6) | -2.2 (0.8) | -1.2 (1.3)

3. Secondary Outcome: Change in Unstimulated Salivary Flow Rate at Wk 4 Post-injection
Description: saliva is collected over 5 minutes and weighed to produce a grams/minute "rate"
Time Frame: baseline vs 4 weeks post-injection
Measure: Mean (Standard Deviation); unit: grams/minute
Arm/Group | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 14
grams/minute | -0.497 (0.38) | -.381 (0.34) | -0.146 (0.14) | -0.052 (0.33)

4. Secondary Outcome: Change in Unstimulated Salivary Flow Rate at Wk 12 Post-injection
Description: saliva collected over 5 minutes and weighed to produce a grams/minute "rate"
Time Frame: baseline vs 12 weeks post-injection
Measure: Mean (Standard Deviation); unit: grams/minute
Arm/Group | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 14
grams/minute | -0.414 (0.37) | -0.166 (0.31) | -0.028 (0.21) | 0.108 (0.35)

ADVERSE EVENTS:
Arm/Group | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 1 | 3
Other Adverse Events (participants affected / at risk) | 2 | 3 | 2 | 1
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Atrial Fibrillation (Cardiac disorders) | 0/14 (0) | 0/12 (0) | 1/13 (1) | 0/15 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0/14 (0) | 0/12 (0) | 0/13 (0) | 1/15 (1)
Rectal Hemmorhage (Gastrointestinal disorders) | 0/14 (0) | 1/12 (1) | 0/13 (0) | 0/15 (0)
Urosepsis (Infections and infestations) | 0/14 (0) | 0/12 (0) | 1/13 (1) | 0/15 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0/14 (0) | 0/12 (0) | 0/13 (0) | 1/15 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0/14 (0) | 0/12 (0) | 0/13 (0) | 1/15 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | 1500U Myobloc | 2500U Myobloc | 3500U Myobloc | Placebo
Dry Mouth (Gastrointestinal disorders) | 1/14 (1) | 2/12 (2) | 1/13 (1) | 0/15 (0)
Breath Odor (Gastrointestinal disorders) | 1/14 (1) | 2/12 (2) | 1/13 (1) | 0/15 (0)
Saliva Altered (Gastrointestinal disorders) | 1/14 (1) | 0/12 (0) | 0/13 (0) | 0/15 (0)
Tongue Coated (Gastrointestinal disorders) | 1/14 (1) | 0/12 (0) | 0/13 (0) | 0/15 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0/14 (0) | 1/12 (1) | 0/13 (0) | 0/15 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 0/12 (0) | 0/13 (0) | 0/15 (0)
Dysgeusia (Nervous system disorders) | 0/14 (0) | 0/12 (0) | 1/13 (1) | 0/15 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0/14 (0) | 0/12 (0) | 0/13 (0) | 1/15 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual investigators may publish results 1 year after the completion of the trial if a multi-center publication has not occurred.